CLINICAL TRIAL: NCT03029520
Title: Termoplastik Kor tekniğini Iki farklı Kanal patı Ile kullanıp Tedavi sonrası Hassasiyet ve kök Ucundan taşma miktarının değerlendirilmesi: Randomize kontrollü Klinik çalışma
Brief Title: Post-Obturation Pain Following the Use of the AH Plus and iRoot SP Sealers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ayfer Atav Ateş, Research assistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAPKOM 4949
Record Dates: First submitted 2017-01-11; First posted 2017-01-24 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Endodontically-Treated Teeth
Keywords: Endodontic Postoperative Pain; iRoot SP Sealer; Randomized Clinical Trial; Herofill carrier-based obturation
MeSH Terms: conditions — Tooth, Nonvital | interventions — Root Canal Obturation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- pain iRoot SP sealer Vital Pulp (Active Comparator): Evaluation of Postoperative pain after root canal obturation with iRoot SP sealer (Innovative BioCeramix Inc., Vancouver, Canada) with patients who has (mandibular premolar/molar) vital pulp.
  Interventions: Other: Root canal obturation with iRoot SP sealer
- pain iRoot SP sealer Devital pulp (Active Comparator): Evaluation of Postoperative pain after root canal obturation with iRoot SP sealer (Innovative BioCeramix Inc., Vancouver, Canada) with patients who has (mandibular premolar/molar) devital pulp.
  Interventions: Other: Root canal obturation with iRoot SP sealer
- pain AHPlus Vital pulp (Active Comparator): Evaluation of Postoperative pain after root canal obturation with AH Plus sealer (Dentsply Maillefer, Ballaigues, Switzerland) with patients who has (mandibular premolar/molar) vital pulp.
  Interventions: Other: Root canal obturation with AH Plus Sealer
- pain AHPlus Devital Pulp (Active Comparator): Evaluation of Postoperative pain after root canal obturation with AH Plus sealer (Dentsply Maillefer, Ballaigues, Switzerland) with patients who has (mandibular premolar/molar) devital pulp.
  Interventions: Other: Root canal obturation with AH Plus Sealer

INTERVENTIONS:
Other: Root canal obturation with iRoot SP sealer — Postoperative pain after root canal obturation with iRoot SP sealer with patients who has (mandibular premolar/molar) vital and devital pulps.
  Arms: pain iRoot SP sealer Devital pulp; pain iRoot SP sealer Vital Pulp
Other: Root canal obturation with AH Plus Sealer — Postoperative pain after root canal obturation with AH Plus sealer with patients who has (mandibular premolar/molar) vital and devital pulps.
  Arms: pain AHPlus Devital Pulp; pain AHPlus Vital pulp

SUMMARY:
The aim of this study was to evaluate and compare postoperative pain and overextension of root canal filling after root canal treatment using a carrier-based obturation system and two different sealers.

In this prospective randomized clinical trial, 160 mandibular premolars and molars in 160 patients were treated. Patients with vital and devital teeth were assigned to four groups using a randomized block design with block sizes of 10 patients each. The groups were composed of devital teeth with periapical lesions treated with iRoot SP sealer, vital teeth treated with iRoot SP sealer, devital teeth with periapical lesions treated with AH Plus sealer, and vital teeth treated with AH Plus sealer. In single visits, a single operator prepared root canals and filled them with sealer using the carrier-based obturation technique. Radiographs were taken and obturation length was recorded. Patients recorded pain scores use of Visual Analogue Scale and frequency of analgesic intake at baseline and 0-6, 6-12, 12-24, and 24-72 h..

DETAILED DESCRIPTION:
This randomized controlled clinical study was conducted to compare the incidence and intensity of post-obturation pain, evaluate the overextension of filling material radiographically, and assess the relationship between pain and analgesic intake in patients with vital and devital teeth undergoing carrier-based obturation with two different sealers (iRoot SP, AH Plus)

ELIGIBILITY:
Inclusion Criteria:

* no systemic diseases
* women were not pregnant or breastfeeding status
* no history of taking analgesics in the previous seven days or other drugs prior to presenting for treatment.
* all selected teeth were mandibular molar or mandibular premolar.

Exclusion Criteria:

* systemic and/or periodontal disease;
* allergy to local anesthetic agents and/or history of intolerance to nonsteroidal anti-inflammatory drugs;
* requirement for antibiotic prophylaxis
* open tooth apex
* pacemaker use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative pain by using VAS scale after obturation with different sealers. | 72 hour

CONTACTS AND LOCATIONS:
Overall Officials: oguz yoldas, professor, Study Chair — vice dean

IPD SHARING:
Plan to Share IPD: Yes
The study will be shared at Turkish Council of Higher education thesis center